CLINICAL TRIAL: NCT05560633
Title: The Feasibility of Nipple-sparing Mastectomy in Combined With Abdominal Free Flap Breast Reconstruction Without Skin Paddles for Flap Monitoring: a Single-center Experience
Brief Title: Nipple-sparing Mastectomy in Combined With Buried Flap Monitoring
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSEC-KY-KS-2021-144
Record Dates: First submitted 2022-09-13; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Breast/Surgery
Keywords: breast cancer; DIEP; ms-TRAM; breast reconstruction; learning curve; nipple spring mastectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
1. Learning curve of ms-Tram and DIEP breast reconstructions surgery are important to guide the training of new surgeon.
2. Buried flap post operative monitoring without implantable doppler was seldom studied, a validated protocol reported.
3. The complication rates of the flap and oncological safety were studied.

DETAILED DESCRIPTION:
Operative time and complication rate are employed to analysis the learning curve of the ms-Tram and DIEP surgery,which is meaningful for the new microsurgeon training.

Buried flap without the implatable doppler is very common condition all over the world, and the complication rate was evaluated as evidence of reliable of the validated monitoring protocol.

Complication rates were considered as different before and after the platue of the learning curve. Within the study of the learning curve, complication rates were reported.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients with age > 18 years
* Received autologous abdominal free-flap breast reconstruction (including muscle-sparing free TRAM or DIEP)

Exclusion Criteria:

* Breast conserving patient
* Implant-based breast reconstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The eligibility of patients for free-TRAM/DIEP was based on the judgement of surgeons, preference of patients, and guideline recommendation as a standard-of-care. For NSM, patients should receive standard-of-care physical examination, ultrasound, mammogram and/or MRI assessment of the involved breast. Patients with clinical involvement of the nipple areola complex (NAC) were excluded
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Total flap failure rate | Through study completion， and average of 2.5 year
  The rate of ms-tram and diep flap were removed from the patients

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li S, Zhang S, Zhang X, Yan J, Wang S, Tan L, Rao N, Chen K, Zhu L. The learning curve of the MS-TRAM/DIEP breast reconstruction by dual-trained breast surgeons. BMC Surg. 2024 Feb 14;24(1):53. doi: 10.1186/s12893-024-02344-z. PMID 38355459